CLINICAL TRIAL: NCT03679351
Title: "Follow Up-Intergroupe Francophone du Myélome 2009" Database Post IFM/DFCI 2009 Study
Brief Title: "FU-IFM2009" Database Post IFM/DFCI 2009 Study
Acronym: DB-FU-IFM2009
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/221
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extension of patient follow-up of the IFM/DFCI 2009 study over a period of 4 years (that is, from 01 December 2016 to 30 November 2020) during which patients will be followed up in the normal course of care and according to the usual care of the centers, with collection of the needed data about twice a year by the investigators

ELIGIBILITY:
Inclusion Criteria:

* Patient randomized in the IFM/DFCI 2009 study.
* Patient still alive must give their non-opposition to the post IFM/DFCI 2009 study data collection until 30 November 2020
* Patient non-opposition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been already randomized in the IFM/DFCI 2009 study
Sampling Method: Non-Probability Sample
Enrollment: 675 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 4 years
  number of deaths

SECONDARY OUTCOMES:
overall long-term survival | 4 years
  number of deaths
secondary primary malignancies | 4 years
  number of secondary primary malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Michel Attal, MD PhD, Principal Investigator — University Hosptial toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France